CLINICAL TRIAL: NCT05141331
Title: Comparison of Piezoelectric Split-crest Technique Versus Expansion Using Hand Driven Ridge Expanders in Treatment of Maxillary Narrow Ridges
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ahmed ashraf abdelreheem (Other)
Responsible Party: Sponsor-Investigator, ahmed ashraf abdelreheem, assistant lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27721
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezoelectric split-crest technique in treatment of Maxillary Narrow Ridges (Experimental): Piezoelectric split-crest technique in treatment of Maxillary Narrow Ridges
  Interventions: Device: piezoelectric
- Hand Driven Ridge Expanders in treatment of Maxillary Narrow Ridges (Active Comparator): Hand Driven Ridge Expanders in treatment of Maxillary Narrow Ridges
  Interventions: Device: piezoelectric

INTERVENTIONS:
Device: piezoelectric — Comparing Piezoelectric split-crest technique versus expansion using Hand Driven Ridge Expanders in treatment of Maxillary Narrow Ridges

SUMMARY:
Comparison of Piezoelectric split-crest technique versus expansion using Hand Driven Ridge Expanders in treatment of Maxillary Narrow Ridges

ELIGIBILITY:
Inclusion Criteria:

* Participants are free from any systemic diseases.
* Participant have missing one or two premolars or molars with sufficient alveolar ridge height and insufficient alveolar ridge buccolingual (BL) width that interfere with conventional straight forward implant placement.
* The minimum BL ridge width included in the study will be 3.5 mm to facilitate ridge splitting and expansion

Exclusion Criteria:

* Patients with residual infections in the edentulous areas.
* Medically compromised groups.
* Smokers and patients with poor oral hygiene.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
bone width | 5 months
  bone width gain in millimeters

SECONDARY OUTCOMES:
implant stability | 5 months
  implant stability measured with periotest

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided